CLINICAL TRIAL: NCT02411370
Title: Correlation Between Respiratory Impairment and Phonemes Alteration in Dystrophinopathy Patients With Respiratory Failure
Acronym: PHONORESPI
Status: Completed | Type: Observational
Sponsor: Centre d'Investigation Clinique et Technologique 805 (Other)
Responsible Party: Sponsor
Other Study IDs: PHONORESPI n°CPP 14079
Record Dates: First submitted 2015-04-03; First posted 2015-04-08 (Estimated); Last update posted 2015-10-15 (Estimated); Status verified 2015-10

CONDITIONS: During the Medical Appointment, the Speech Therapist Will Perform Phonetic Tests

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

INTERVENTIONS:
Behavioral: phonetic tests

SUMMARY:
Communication is essential for patients quality of life because it impact on patients care quality. Neuromuscular diseases, caracterised by motor damages, hinder non-verbal communication of the patient. Therefore, speech must to be functional.

However, correlation between respiratory failure and voice quality is not very well known. The aim of the study is to search a link between respiratory failure and speech impairment in patients with neuromuscular diseases.

ELIGIBILITY:
Inclusion Criteria:

* Respiratory autonomy at least 1 hour per day
* Stable patient during the study
* Patient with education at least up to secondary school

Exclusion Criteria:

* Refusal to participate
* Inability to cooperate
* Tracheostomized patients
* Mechanic ventilation - dependant patients
* Respiratory autonomy lower than 1 hour per day
* Patients with hemodynamic instabillity
* Patient insured under the French social security system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Dystrophinopathy patients with limitive respiratory failure.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2015-02; Primary Completion 2015-06 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Intelligibility phonetic test | 5 minutes
Number and nature of altered phonemes | 5 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Raymond-Poincaré, Garches, Hauts-de-Seine, France